CLINICAL TRIAL: NCT06403592
Title: The Effect of a Laryngeal Mask Airway on Optic Nerve Sheath Diameter
Acronym: ONSD laryngeal
Status: Recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Iscander M Maissan, Dr., Erasmus Medical Center
Other Study IDs: ONSD laryngeal
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Intracranial Pressure Increase
Keywords: Laryngeal airway mask; Optic Nerve sheath Diameter; Intracranial Pressure
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational cohort: ASA I-II patients scheduled for surgery under general anesthesia with a laryngeal airway mask
  Interventions: Other: optic nerve sheath diamater

INTERVENTIONS:
Other: optic nerve sheath diamater — Measurement of optic nerve sheath diameter

SUMMARY:
The goal of this observational trial is to study the effect of a laryngeal airway mask on the optic nerve sheath diameter, as a surrogate for intracranial pressure.

The optic nerve sheath diameter of participants will be measured under general anesthesia, before, during and after insertion of a laryngeal airway mask.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, a subject must meet all of the following criteria: aged 18 years or older, ASA I or ASA II, scheduled for elective surgery under general anesthesia, with a planned duration of > 30 minutes, that can be routinely performed with a LMA.

Exclusion Criteria:

* Scheduled for head or neck surgery
* Scheduled for neurosurgery
* Scheduled for laparoscopic or thorascoscopic procedures
* Scheduled for procedures that require Trendelenburg or anti-Trendelenburg positioning
* Neurological disorders
* Glaucoma
* History of bilateral eye related trauma
* Intellectual disability

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ASA I-II patients scheduled for surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Effect of insertion of a laryngeal airway mask on optic nerve sheath diameter | During surgery

SECONDARY OUTCOMES:
Effect of laryngeal ariway mask after insertion on optic nerve sheath diameter | During surgery
Effect of layngeal airway mask on optic nerve sheath diameter interna vs optic nerve sheath diameter externa | During surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medisch Centrum, Rotterdam, Netherlands